CLINICAL TRIAL: NCT01656941
Title: The GECHO Trial: Genetic Determinants of Congenital Heart Disease Outcomes
Brief Title: Genetic Determinants of Congenital Heart Disease Outcomes
Acronym: GECHO
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Royal Children's Hospital (Other); Medical University of South Carolina (Other); Emory University (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Mark Russell, Professor of Pediatric Cardiology and Professor of Pediatrics, University of Michigan
Other Study IDs: GECHO
Record Dates: First submitted 2012-07-19; First posted 2012-08-03 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Congenital Heart Disease; Hypoplastic Left Heart Syndrome; Hypoplastic Right Heart Syndrome; d-Transposition of the Great Arteries
Keywords: neonate; congenital heart disease; single ventricle cardiac disease; hypoplastic left heart syndrome; hypoplastic right heart syndrome; d-Transposition of the Great Arteries
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be frozen and stored until DNA can be isolated. Eventually, isolated DNA samples will be frozen and stored in a biorepository.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- d-Transposition of the Great Arteries: Neonates with d-transposition of the great arteries (dTGA) undergoing the arterial switch operation with cardiopulmonary bypass
- Single ventricle cardiac disease: Neonates with single ventricle cardiac disease (SVCD) undergoing stage I surgical palliation (Norwood) with cardiopulmonary bypass

SUMMARY:
The purpose of this study is to examine the role of genetic variation in the oxidative stress response on critical perioperative and short-term outcomes after neonatal heart surgery. The goals will be to determine 1) if the oxidative stress pathway is an important one for therapeutic intervention in neonates with severe congenital heart defects and 2) if variants in the oxidative response pathway can be used to identify patients at increased risk for adverse outcomes.

DETAILED DESCRIPTION:
For physicians caring for children with congenital cardiac defects, perhaps the greatest challenge is to improve the survival and functional outcomes of patients with severe defects requiring surgical repair or palliation in the first month of life. These cardiac defects can be associated with 5 year mortality rates of up to 30% with significant disabilities in many of the survivors. As with every medical condition, patient outcomes depend on the complex interaction of the disease process, the medical and surgical interventions to treat the disease, and the inherent capacity of the patient to respond to both the disease and its treatment.

For patients with severe cardiac defects, the greatest risk for morbidity and mortality occurs during and shortly after their neonatal surgical repair. During surgery to repair severe cardiac defects, the body is cooled and the heart is stopped. In many cases, blood flow to the vital organs is interrupted or restricted for a significant period of time while the aortic arch is reconstructed. This process places profound stress on the patient's capacity to tolerate these insults without sustaining irreversible injury to tissues such as the heart, brain, and kidneys. That there is such a wide range of outcomes after this surgery, even between patients with similar clinical features, suggests that there are important individual differences in patients' abilities to respond to this stress that is determined by differences in their genetic traits.

The importance of the interaction between the controlled trauma of the surgical environment and a patient's genetic background in determining patient outcomes has led to the new discipline of "peri-operative genomics." In this study, we will examine the contribution of gene-environment interactions to perioperative and short-term outcomes in neonates with severe congenital cardiac defects.

ELIGIBILITY:
Inclusion Criteria:

* d-transposition of the great arteries or single ventricle cardiac disease
* Less than or equal to 30 days of age
* Planned arterial switch operation or stage I surgical palliation (Norwood)with aortic arch reconstruction

Exclusion Criteria:

* Known trisomy 13, 18, or 21
* Any major non-cardiac anomaly that precludes the patient from cardiac surgery

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with d-transposition of the great arteries undergoing the arterial switch procedure and neonates with single ventricle cardiac disease undergoing stage I surgical palliation at the University of Michigan or other collaborating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-03; Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Contribution of genetic variation in oxidative stress management to differences in short term outcomes after repair for severe cardiac disease in the neonatal period | Duration of initial perioperative hospitalization (~2-4 weeks)
  Genotyping will be performed on 10 variants in the oxidative stress response pathway and we will combine risk genotypes in order to evaluate the cumulative effect of both detrimental and beneficial alleles on post-operative outcomes.
  Composite short term outcome measure includes:
  ICU length of stay (days) Time to initial extubation (hours) Cardiac arrest or ECMO support (Y/N) Delayed sternal closure (Y/N) Serious adverse event (Y/N) Greater than 1 serious adverse event (Y/N)

SECONDARY OUTCOMES:
Contribution of genetic variation in oxidative stress management to differences in interstage mortality and pre-Stage II cardiovascular function in patients with single ventricle cardiac disease | Interval from hospital discharge following stage I surgical palliation until hospital admission for stage II surgical palliation (~4-6 months of age)
  Composite outcome
  * Growth parameters (height, weight, head circumference)
  * AV valve insufficiency (By echocardiogram and cardiac catheterization) , Ventricular function (ejection fraction by echocardiogram and by cardiac catheterization), Central venous pressure and ventricular end diastolic pressure (by catheterization), Interstage Death (Y/N).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole S Wilder, MD, Principal Investigator — University of Michigan; Mark W Russell, MD, Principal Investigator — University of Michigan
Locations (5):
- United States (4):
  - Emory University, Atlanta, Georgia
  - C.S. Mott Children's Hospital, University of Michigan Health System, Ann Arbor, Michigan
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Royal Children's Hospial Melbourne, Melbourne, Victoria, Australia